CLINICAL TRIAL: NCT05778084
Title: Effect of Empagliflozin on NT-Pro Brain Natriuretic Peptide in Heart Failure Patients With Reduced Ejection Fraction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0107427
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Empagliflozin; Heart failure with reduced ejection fraction; Nt-proBNP
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Open labelled interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart failure patients with reduced and mildly reduced ejection fraction (Other): * One paired test group described as Heart Failure patients with reduced and mildly reduced ejection fraction are indicated for Empagliflozin.
  * Blood samples will be collected as a baseline before Empagliflozin administration to test for N-terminal Pro-B-type Natriuretic Peptide,
  * Followed by administration of empagliflozin for 6 months.
  * Then retest the N-terminal Pro-B-type Natriuretic Peptide after 6 months.
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Blood samples will be collected as a baseline to test for N-terminal Pro-B-type Natriuretic Peptide, followed by administration of empagliflozin for 6 months, and then another blood samples will be collected after 6 months.

SUMMARY:
This study aims to evaluate the relationship between NT-proBNP and empagliflozin effects in patients with chronic heart failure with mildly reduced ejection fraction (HFmrEF 41-49%) and reduced ejection fraction (HFrEF ≤40%) whether diabetic or non-diabetic patients.

DETAILED DESCRIPTION:
1. Ethical Committee approval has been obtained from ethics committee of Faculty of Medicine, Alexandria University.
2. Assigning an informed consent for agreement of participation should be taken by all participants in this clinical study.
3. Heart failure patients with reduced and mildly reduced ejection fraction will be recruited from Alexandria Main University Hospital (AMUH), private hospitals and clinics.
4. A Blood sample will be collected from 60 patients as baseline to test for N-terminal Pro-B-type Natriuretic Peptide.
5. The same 60 patients will take Empagliflozin for 6 months.
6. Another blood sample will be taken from the same 60 patients to test the effect on N-terminal Pro-B-type Natriuretic Peptide after Empagliflozin administration.
7. The appropriate statistical test will be hold according to study design and parameters to evaluate the significant results.
8. Results conclusion discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure with mildly reduced ejection fraction (41-49%) and reduced ejection fraction (≤40%)
* 18-70 years
* Not receiving empagliflozin or any SGLT2 inhibitor
* Elevated plasma NT-proBNP (≥125 pg/ml)
* eGFR ≥ 20 ml/min/1.73m2

Exclusion Criteria:

* Acute Coronary Syndrome (ACS)
* Pulmonary embolism
* Myocarditis
* Valvular heart disease
* Hypertrophic or restrictive cardiomyopathy
* Congenital heart disease
* Pulmonary hypertension
* Surgical procedures involving the heart
* Heart contusion
* Cardioversion, Implantable Cardioverter Defibrillator (ICD) shock
* Patients receiving digoxin
* Advanced age (>70years)
* Ischemic stroke
* Chronic Obstructive Pulmonary Disease
* Subarachnoid haemorrhage
* Severe infection (including pneumonia and sepsis)
* Anemia
* Renal dysfunction (eGFR <20ml/min/1.73m2)
* Liver dysfunction (mainly liver cirrhosis with ascites- Child Pugh B & C)
* Severe burns
* Paraneoplastic syndrome
* Severe metabolic and hormone abnormalities (e.g thyrotoxicosis, diabetic ketosis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
NT-ProBNP | 6 months
  Measuring of serum N-terminal Pro-B-type Natriuretic Peptide at baseline and after 6 months

SECONDARY OUTCOMES:
Hemoglobin level g/dl | 6 months
  Measuring hemoglobin level at baseline and after 6 months
Leukocytes count | 6 months
  Measuring Leukocytes count at baseline and after 6 months
Sodium level mg/dl | 6 months
  Measuring serum sodium level at baseline and after 6 months
Potassium level mg/dl | 6 months
  Measuring serum potassium level at baseline and after 6 months
Serum Creatinine | 6 months
  Measuring serum creatinine level at baseline and after 6 months
Ejection Fraction | 6 months
  Measuring Ejection Fraction at baseline and after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No